CLINICAL TRIAL: NCT02105480
Title: Automated Algorithm Based Analysis of Phonocardiograms of Newborns
Status: Completed | Type: Observational
Sponsor: CSD Labs GmbH (Other)
Responsible Party: Sponsor
Other Study IDs: GRZ02 (AAAPN)
Record Dates: First submitted 2014-03-31; First posted 2014-04-07 (Estimated); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: Heart Murmurs; Mitral Valve Prolapse; Systolic Murmurs
Keywords: Computer aided auscultation (CAA); Phonocardiogram analysis; Murmur detection; Heart auscultation
MeSH Terms: conditions — Heart Murmurs; Mitral Valve Prolapse; Systolic Murmurs

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Computer aided auscultation (CAA)
  Other Names: Phonocardiogram analysis; Automated heart murmur classification; Murmur screening

SUMMARY:
The purpose of this double-blind pivotal clinical utility study is to determine on a large patient population whether heart murmurs can be reliably detected with high sensitivity and specificity using a locked, automated algorithm-based phonocardiogram analysis (also referred to as computer aided auscultation (CAA)).

Each patient is auscultated and diagnosed independently by a medical specialist. Additionally, for each patient, an echocardiogram is performed as the gold-standard for determining heart pathologies. The CAA results are compared to the findings of the medical professionals as well as to the echocardiogram findings.

Hypothesis: The specific (locked) CAA algorithms used in this study are able to automatically diagnose pathological heart murmurs in premature babies and newborns with at least the same accuracy as experienced medical specialists.

DETAILED DESCRIPTION:
The following registry procedures and quality factors have been implemented:

* Quality assurance plan, including

  * data validation
  * proper registration procedures
  * regular site monitoring
  * regular auditing
* Data checks to compare data entered into the registry against predefined rules for range or consistency with other data fields in the registry.
* Source data verification to assess the accuracy, completeness, or representativeness of registry data by comparing the data to external data sources (medical records and paper case report forms).
* Standard Operating Procedures to address registry operations and analysis activities, such as patient recruitment, data collection, data management, data analysis, reporting for adverse events, and change management.
* Sample size assessment to specify the number of participants or participant years necessary to demonstrate an effect.
* Statistical analysis plan describing the analytical principles and statistical techniques to be employed in order to address the primary and secondary objectives, as specified in the study protocol or plan.
* Plan for missing data to address situations where variables are reported as missing, unavailable, "non-reported," uninterpretable, or considered missing because of data inconsistency or out-of-range results.

ELIGIBILITY:
Inclusion Criteria:

* any premature baby or newborn
* parental approval for study participation

Exclusion Criteria:

* none

Ages: 1 Minute to 5 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Premature babies and newborns stationed at the department of neonatology
Sampling Method: Non-Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2016-01-25 (Actual); Study Completion 2017-01-18 (Actual)

PRIMARY OUTCOMES:
Number of correctly diagnosed heart murmurs through locked, independent algorithm based auscultation and traditional stethoscope based auscultation by medical experts | 2 years (expected)
  Each patient is screened and diagnosed regarding a potential heart murmur by a medical expert through standard stethoscope based auscultation. Heart sounds are recorded using an electronic stethoscope and analyzed and diagnosed independently (with no external input) by a locked algorithm. A final diagnoses for each patient is made by a medical expert by performing an echocardiogram, the gold standard method for heart murmur detection. The diagnoses of both the medical expert and the algorithm are finally compared to the echocardiogram based diagnosis (after completion of patient recruitment).

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Pichler, MD, Principal Investigator — Medical University of Graz
Locations (1):
- University Hospital, Graz, Styria, Austria